CLINICAL TRIAL: NCT04384874
Title: SSC6 Versus Silbernagel Rehabilitation Program in Patients With Chronic Mid-portion Achilles Tendinopathy: A Randomised Control Trial
Brief Title: A Novel Multi-factorial Criteria-based Rehabilitation Program for Chronic Mid-portion Achilles Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sports Surgery Clinic, Santry, Dublin (Other)
Responsible Party: Principal Investigator, Dr Neil Welch ASCC, Head of lab services and research, Sports Surgery Clinic, Santry, Dublin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSC-Achilles-001
Record Dates: First submitted 2020-04-23; First posted 2020-05-12 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Achilles Tendinopathy
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silbernagel combined concentric-eccentric program (Active Comparator): A graduated rehabilitation program using exercises with concentric and eccentric contractions and progressing to plyometric training. The exercises are performed daily with progression guided by pain symptoms. There is no specificity in prescribed exercise loading.
  Interventions: Other: Exercise therapy
- SSC6 (Experimental): A multi-stage rehabilitation program with focus on strength and reactive strength targets, as well as running gait re-training. These exercises will be initially carried out 3 days per week for the first 6 weeks with specific load targets prescribed.
  Interventions: Other: Exercise therapy

INTERVENTIONS:
Other: Exercise therapy — A 12 week multi-stage exercise rehabilitation program

SUMMARY:
Sixty physically active patients (aged 18-45) with chronic mid-portion Achilles tendinopathy will be recruited to take part in the study. The patients will be diagnosed by a sports medicine doctor and an MRI scan and will be experiencing palpable Achilles pain at the time of inclusion. The patients will be randomized into either a group performing the Silbernagel combined concentric-eccentric program, or a group performing a novel multi-phase program with specific outcome measures. The study will assess the patients calf strength, reactive strength and running biomechanics at baseline, week's 6 and 12 of a rehabilitation program and be available for a 6 month, 12 month and 2 year follow-up interview. The VISA-A questionnaire will be the primary outcome measure and will be completed at each testing and follow-up session.

DETAILED DESCRIPTION:
Achilles tendinopathy is an overuse injury commonly seen in sports and physical activities that involve running, jumping and hopping. Patients with Achilles tendinopathy experience pain, morning stiffness and reduced ability to exercise. This condition can last for several years in some cases.

Exercise therapy in the form of resistance training has been demonstrated to be the most effective rehabilitation tool to reduce pain and increase function in patients with Achilles tendinopathy. Patients often experience clinical improvements before any meaningful structural changes on MRI or ultrasound imaging are observed. Returning athletes back to competitive sport requires a progressive loading program to enable them to tolerate high stretch-shortening cycle loads appropriate to the demands of their sport.

The SSC6 rehabilitation program is a six-stage pathway with a focus on strength development of the local muscle-tendon unit and the kinetic chain, the development of power and kinetic strength, running biomechanics and running load modification. The progression through each phase is guided by objective outcome criteria based on pain and function, strength and performance tests and achieving individualised resistance load targets. The strength and power exercises are performed at high intensity three days per week with 48 hours recovery. The Silbernagel program is a four-phase involves a daily exercise program of lower intensity with progression through each phase guided by symptoms and function.

This study will compare the effectiveness of a comprehensive Achilles tendinopathy rehabilitation program with progression criteria with a common Achilles tendinopathy rehabilitation program. Sixty recreationally-active subjects aged between 18-45 years who meet the inclusion criteria, will be recruited to partake in this study. The subjects will be randomly assigned to one of two groups where they will undergo a multi-phase rehabilitation program. Data will be collected at baseline, 6 weeks and 12 weeks, to monitor pain and functional response, biomechanical and structural changes. At 6, 12 and 24 months following the commencement of the rehabilitation program, patients will be required to complete a follow-up questionnaire to monitor progress and any re-injury incidence that may have occurred.

The following testing protocols will be performed:

1. VISA-A Questionnaire The VISA-A questionnaire has been shown to be a valid, reliable and easy to use outcome measure tool for intervention studies on Achilles tendinopathy. It consists of eight questions regarding pain and function during both daily living and sporting activities. The overall score is between 0-100 where higher scores represent reduced pain and improved function. An improvement of 21 points between 2 and 12 weeks of a rehabilitation program have been typically observed. The difference in VISA-A score between both training protocols from baseline testing to the outcome testing at 6 weeks, 12 weeks, 6 and 12 months; will formulate the primary outcome measure for this study.
2. Ankle isokinetic testing Achilles tendinopathy has been associated with reduced plantar flexor strength. Isokinetic testing is commonly used to measure plantarflexor peak torque. The subjects will perform 2 isokinetic tests. In the first test the subjects will lie in a prone position in an isokinetic dynamometer with full knee extension and the foot securely strapped to a pedal a neutral ankle position (tibia perpendicular to the sole of the foot). The centre of rotation of the ankle axis will be aligned with the dynamometer. Subjects will be asked to perform a warm-up involving 5 sub maximal concentric plantarflexion and dorsiflexion contractions between 60-100% of their self-perceived MVC. The subjects will then be required to produce a maximal plantarflexion force 5 repetitions for 2 sets with a 1 minute rest between sets. In the second test the subjects will lie in supine position with the knee flexed to 80º in order to specifically test the peak torque of the soleus. The same warm-up protocol and sets and repetitions as the previous test will apply. Both tests will use a speed of 60º per second and operate through an ankle range of between 30º plantarflexion and 20º dorsiflexion.
3. Running biomechanics Altered running biomechanics and muscle recruitment strategies have been highlighted in runners with Achilles tendinopathy. The subjects will be asked to run on the treadmill at a self-selected sub maximal speed. Using 3D motion analysis (Run 3D, Oxford, United Kingdom), a number of biomechanical variables will be measured. These include: vertical and leg stiffness, contact time, flight time, stride length, stride frequency and joint angular displacements from initial contact to mid stance phase.
4. Hop testing Achilles tendon material properties contribute to stretch shortening cycle performance during hopping tasks. Reduced tendon mechanical properties, plantar flexor muscle rate of force development and deficits on a single leg horizontal hop have previously been observed in patients with Achilles tendinopathy. Jump height, ground contact time and reactive strength index (RSI) will be measured using a double and single leg drop jump. Vertical, leg and ankle joint stiffness will be calculated using a novel single leg hurdle hop test. A pilot study has previously been carried out on 10 healthy subjects prior to the commencement of the Achilles RCT study. Good to excellent reliability was found for of vertical stiffness, contact time, ground reaction force, hop distance and rebound distance and 3 trials were sufficient to obtain a true measure of performance across most variables.
5. Subjective questionnaire After the completion of the rehabilitation program patients will be ask to provide feedback on the prescribed program and will complete a training diary where compliance and adherence to the program will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with mid-portion Achilles Tendinopathy by a sports medicine physician
* Have experienced symptoms for more than 3 months and less than 3 years
* Aged between 18-45 years,
* Regularly perform running-based exercise more than twice per week

Exclusion Criteria:

* Have a co-existing lower limb injury.
* Have had another running-related injury in the previous 12 months.
* Have had an Achilles injection in the past 6 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Change in VISA-A Questionnaire score | This will be assessed at week 6 and 12, as well as 6, 12 and 24 month follow-ups
  This is a measure of pain and lower limb function associated with Achilles tendinopathy and a primary outcome measure will be the change in VISA-A questionnaire at various time points during the 12 week intervention and in the long-term follow-ups. A change of 20 points is typically observed after a rehabilitation program, while a 10 point increase is accepted as being clinically meaningful.

SECONDARY OUTCOMES:
Plantar flexor strength | This will be carried out at week 0, 6 and 12
  Measured using isokinetic dynamometry to determine plantar flexor peak torque relative to bodyweight (Nm/kg) with 2 test protocols.
Running biomechanics | This will be carried out at week 0, 6 and 12
  Using 3D motion analysis (Run 3D, Oxford, United Kingdom) a number of kinematic and spatiotemporal variables will be measured: contact time, flight time, stride length, stride frequency and joint angular displacements from initial contact to mid stance phase. Spring mass model characteristics and especially lower limb stiffness will be calculated using a validated equitation based on running speed, contact time, body mass and leg length dimensions. After a brief warm-up, the subject will be asked to run at a speed they feel that they could sustain for a 30 minute steady effort and data will be captured for 30 seconds. The running speed selected by the subject at baseline testing will be repeated for the two subsequent testing sessions.
Lower limb reactive strength | This will be carried out at week 6 and 12
  Patients will be asked to perform a double and single leg vertical drop jump and a single leg horizontal rebound task to assess lower limb biomechanics and reactive strength qualities.

CONTACTS AND LOCATIONS:
Locations (1):
- Sports Surgery Clinic, Dublin, Leinster, Ireland

REFERENCES:
- [Derived] Griffin C, Daniels K, Hill C, Franklyn-Miller A, Morin JB. A criteria-based rehabilitation program for chronic mid-portion Achilles tendinopathy: study protocol for a randomised controlled trial. BMC Musculoskelet Disord. 2021 Aug 14;22(1):695. doi: 10.1186/s12891-021-04553-6. PMID 34391384